CLINICAL TRIAL: NCT06486805
Title: The Effect of N-Acetylcysteine on Liver Functions After Mitral Valve Replacement: A Randomized Controlled Trial
Brief Title: N-Acetyl Cysteine Effect on Liver Function After Mitral Valve Replacement
Acronym: NAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohamed Elhaddad, Assisstent professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-66-2017
Record Dates: First submitted 2024-06-21; First posted 2024-07-05 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-06

CONDITIONS: Oxidative Stress; Liver Dysfunction
Keywords: MDA; liver function; N-acetylcystien
MeSH Terms: conditions — Liver Diseases | interventions — Acetylcysteine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: quadrible blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Placebo Comparator): received the same volume of normal saline as placebo
  Interventions: Other: normal saline
- NAC (Active Comparator): received 150 mg/kg NAC in 200 ml of 5% glucose over 15 min through the central line after induction of anesthesia and intubation followed by 50 mg/kg of NAC in 500 ml of 5% glucose over 4 h
  Interventions: Drug: N acetyl cysteine

INTERVENTIONS:
Drug: N acetyl cysteine — N-acetylcysteine (NAC) is a small molecule containing a thiol (sulfhydryl-containing) group, which has antioxidant properties and is freely filterable, thus making it readily accessible to the intracellular compartment
  Other Names: NAC
  Arms: NAC
Other: normal saline — the same volume of normal saline
  Other Names: placebo
  Arms: control

SUMMARY:
This study aimed at the impact of the N-acetyl cysteine on the improvement of liver function subsequently on-pum mitral valve replacement. Following a clinical trial design, 54 candidates of on-pump MVR, aged 18 to 70 years, with normal liver and renal function were selected. The candidates were randomly divided into intervention: IV150 mg/ kg N-acetyl cysteine over 15 min, and control groups (normal saline as placebo) (n = 27 in each group).

DETAILED DESCRIPTION:
In a randomized controlled prospective study conducted in a teaching hospital, after approval by the ethics committee and informed consent, 54 candidates for on-pump MVR, aged 18 to 70 years, with normal liver and renal function, were selected. The candidates were randomly divided into intervention: IV 150 mg/ kg N-acetyl cysteine over 15 min then 50 mg/kg over 4 hrs for 3 days, and control groups (normal saline as placebo) (n = 27 in each group).and we will assess the effect of NAC on intra-operative hemodynamics and post-operative its protective rule against oxidative stress and liver dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70 years
* Both sexes
* Patients undergoing on-pump elective MVR with cold cardioplegia.

Exclusion Criteria:

* Patient refusal.
* Allergy to any of the study medications.
* Emergency procedures.
* systolic dysfunction, left ventricular ejection fraction <40%.
* Pre-existing hepatic dysfunction, which is defined as an increase in liver enzymes AST and ALT >10 times the baseline.
* chronic use of drugs affecting liver functions, e.g., NSAIDs, steroids, and anticonvulsants.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Malondialdahyde (MDA) | Postoperative day one
  MDA is a marker of oxidative stress and one of the end-products of lipid peroxidation. MDA level reflects the degree of lipid peroxidation.

SECONDARY OUTCOMES:
MDA | preoperative and second postoperative day
  MDA is a marker of oxidative stress and one of the end-products of lipid peroxidation. MDA level reflects the degree of lipid peroxidation.
liver function tests | preoperative ,first ,and,second post operative days
  ALT,AST,Bilirubin
hemodunamics | intraoperative
  MAP, HR
extubation time | postoperative 24 hr.
  time needed for extubation
tissue perfusion | preoperative ,first ,and,second post operative days
  Lactate

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralainy Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No